CLINICAL TRIAL: NCT01788059
Title: The Efficacy of Mesenchymal Stem Cells for Stimulate the Union in Treatment of Non-united Tibial and Femoral Fractures in Shahid Kamyab Hospital
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emdadi Kamyab Hospital (Other)
Responsible Party: Principal Investigator, mohammad taghi peivandi, MD, Emdadi Kamyab Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 900939
Record Dates: First submitted 2013-01-17; First posted 2013-02-11 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Nonunion Fracture
Keywords: nonunion; mesenchymal stem cell; long bone
MeSH Terms: conditions — Fractures, Ununited

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mesenchymal stem cell (Experimental): stem cells drived from iliac bone marrow with centrifuge and ficoll method then inject to non union site 2-3 ml with approximately 40 X 10E6 Mesenchymal Stem Cells (MSC) will be injected in the nonunion site of the bone fracture under fluoroscopic gide and general or spinal anesthesia as deemed appropriate by the anesthetist.
  Interventions: Other: injection the mesenchymal stem cell in non union site

INTERVENTIONS:
Other: injection the mesenchymal stem cell in non union site

SUMMARY:
Because the rate of non union of long bone in lower extremities specially in tibia in this two last decade due to malnutrition and smoking and other risk factors was increased, so many patient in our country suffer from non union on the other hand it seems that the use of the mesenchymal stem cells can irritate the union rate. Therefore the investigators decide to inject the mesenchymal stem cell derived from iliac bone marrow after centrifuge with ficoll procedure to non union site in patient that are resistant to other treatment. Then the investigators will follow the patient with monthly radiography and evaluate the callus volume and clinical union and any side effect of this treatment.clinical union consider to relief pain in non union site and be stable in examination.

ELIGIBILITY:
Inclusion Criteria:

* Every patient with non union in the site of long bone fracture
* Age more than 18 and under 60 years old
* Fracture having no radiological callus after 6 months and absence of any hypertrophic bone reaction.
* No infection in site of surgery
* Be able and willing to participate in the study
* Written informed consent

Exclusion Criteria:

* Evidence of malignancy
* Pregnancy or breastfeeding
* Patient positive by serology or PCR for HIV, hepatitis B or C infection the patient with Accompanied fracture such as hip fracture that could not weight bearing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
clinical and radiological union at 1 month to 6 months | 6 months
  patients receiving Mesenchymal Stem Cells that develop a partial or complete callus at 1, 2, 3, 4 ,5 and 6 months evaluate with standard X-rays

SECONDARY OUTCOMES:
•Safety of Mesenchymal Stem Cells injection in nonunion fractures. Follow-up for revealing any significant immediate or late adverse effects. | 12 months
Incidence of adverse events in patients (e.g infection , malignancy , ...) Adverse events will be continuously monitored | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: mohammad taghi peivandi, MD, Principal Investigator — Emdadi Kamyab Hospital
Locations (1):
- Emdai Kamyab Hospital, Mashhad, Khorasan, Iran